CLINICAL TRIAL: NCT07087691
Title: Pilot Post-Marketing Study on the Efficacy of OneMark in Identifying Breast Cancer For Surgery and Over Time in High and Low Density Breast Tissue
Brief Title: Efficacy of OneMark Device in Identifying Breast Cancer for Surgery and Surveillance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: View Point Medical (Unknown)
Responsible Party: Principal Investigator, Sara Grossi, Assistant Professor of Clinical Surgery, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 812244
Record Dates: First submitted 2025-07-08; First posted 2025-07-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; suspicion of breast cancer; fiducial; visualization device
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Breast cancer surgical resection (Experimental): Participants with stage T1/T2 breast cancer visible by ultrasound and scheduled for breast cancer surgical resection.
  Interventions: Device: OneMark device
- Breast cancer surveillance (Experimental): Participants with Breast Imaging Reporting and Data System (BI-RADS) category 4 or 5 on screening mammogram, with lesions visible by ultrasound, and entered in a surveillance program.
  Interventions: Device: OneMark device

INTERVENTIONS:
Device: OneMark device — The OneMark device system consists of a tumor marker preloaded in a delivery system, a handheld probe, and a display console.
  The OneMark marker is a metal clip with microparticles embedded in gelatin forming a hydrogel pellet. The pellet is implanted with a preloaded injector percutaneously in soft tissues, such as breast or lymph nodes, to mark a biopsy site or tissue intended for surgical removal. It can be used as a fiducial implant post-biopsy for future identification or monitoring of the tissue, and as an intra-operative localization mark. The microparticles of OneMark marker can be detected by Doppler ultrasound, magnetic resonance imaging (MRI), radiography, and OneMark Detector. During surgery, the OneMark marker may be removed with the target tissue. If patients do not require surgery, the OneMark marker can be left in place.

SUMMARY:
The goal of this research is to study a localization device for breast cancer called OneMark. This device will be studied in breast cancer surgery and during surveillance in patients being monitored for breast cancer.

The main questions the study aims to answer are:

Can surgeons visualize the OneMark device during breast cancer surgery better than a standard of care visualization device?

Can radiologists visualize the OneMark device over time during breast cancer surveillance in patients with low or high density breast tissue?

Participants will undergo breast cancer surgery or surveillance as required for their regular care. For patients undergoing surgery, the device will be implanted ahead of surgery. For patients in surveillance, the device will be implanted during biopsy and visibility of the device will be assessed by radiologists after 1, 3, and 6 months, and optionally after 12 months.

Surgeons will complete a questionnaire at every surgery on the visibility of the OneMark device and the standard of care visualization device. Radiologists will complete a questionnaire after 1, 3, 6 months (and optionally after 12 months) after implantations in the patients in the surveillance program.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-site study to evaluate the OneMark visualization device in 2 patient populations: patients with breast cancer undergoing resection surgery, and patient at high risk of breast cancer in a surveillance program. In addition, the study enrolls 2 physician populations: surgeons and radiologists specialized in breast cancer.

In the surgery cohort, the investigators will compare the OneMark device to the standard of care wireless localization system, SAVI SCOUT. The visibility of the two devices will be evaluated before, during, and after surgery (ex vivo).

In the surveillance cohort, the investigators will evaluate the detectability over time of the OneMark device placed as fiducial during breast biopsy in patients with low or high density breast tissue. If participants in the surveillance group will require surgery during the study, the surgeons can opt to place a SAVI SCOUT marker and will evaluate the visibility of both devices like in the cohort described above.

We hypothesize that the OneMark device has superior intra-operative visibility compared to the SAVI SCOUT system for detection of breast cancer for surgical resection. We also hypothesize that, when the OneMark device is used as fiducial during surveillance, it will be visible over time.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Age ≥ 18 years.
* In good general health as evidenced by medical history.
* Deemed able to undergo general anesthesia for surgical resection.
* For individuals who are capable of menstruating: must be post-menopausal, defined as no menses in the 12 months before enrollment or age > 60 years. No additional requirements - besides the age requirement in inclusion criterion # 3 - are needed for individuals who are not capable of menstruating.

For surgery cohort only:

* Male and female patients with stage T1/T2 breast cancer visible by ultrasound.

For surveillance cohort only:

* Male and female patients with abnormal mammogram Breast Imaging Reporting and Data System (BI-RADS) category 4 or 5.
* Ultrasound visible unifocal breast tumor < 5 cm in diameter.
* Low density tissue by mammogram either category A (fatty replaced) or category B (scattered densities); or high density tissue by mammogram either category C (heterogeneously dense) or category D (extremely dense).

Exclusion Criteria:

* Pregnancy or lactation.
* Known allergic reactions to components of OneMark System or SAVI SCOUT.
* Feverish illness within 7 days of placement of the device.
* Previous treatment with another investigational drug or other intervention within 1 month of enrollment.
* Previous use of neoadjuvant chemotherapy within 6 months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of visibility rankings of OneMark marker and SAVI SCOUT | At time of surgery
  Visibility rankings of OneMark marker and SAVI SCOUT on a 4-point scale. Grade 0: no visibility; Grade 1: uncertain visibility; Grade 2: some visibility; Grade 3: definite visibility.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Grossi, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No